CLINICAL TRIAL: NCT05744102
Title: Evaluation of Advanced and New MRI Techniques to Improve Patient Diagnosis
Brief Title: Improve MRI Diagnosis
Acronym: DIAGIRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220840; 2022-A01358-35 (Other: IDRCB)
Record Dates: First submitted 2023-01-23; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: New MRI Techniques
Keywords: Advanced MRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients having MRI planned at Paul Brousse Hospital (Other): Evaluate new MRI sequences on a population of patients undergoing MRI as part of their usual care
  Interventions: Diagnostic Test: MRI Image

INTERVENTIONS:
Diagnostic Test: MRI Image — MRI sequences

SUMMARY:
The main objective of the research is to compare by two blind evaluators new MRI techniques with routinely used sequences.

DETAILED DESCRIPTION:
"The main evaluation criterion will be the choice of the two (or three) evaluators as to the best sequence between the new sequence and the standard sequence.

The decision criterion for considering a new sequence as superior to the standard sequence will be based on two measures:

1. The proportion of patients for whom the new sequence was preferred, which must be greater than or equal to 75%;
2. Inter-observer agreement (Cohen's Kappa coefficient), which must be greater than or equal to 0.8; When these two criteria are met, the new sequence will be considered superior to the standard sequence"

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who signed a consent to participate in the study
* Affiliated patient or beneficiary of a social security scheme
* Patient having an MRI scheduled as part of their care pathway
* Absence of prohibition of participation in another research

Exclusion Criteria:

* Patients under guardianship or curators
* Pregnant or breastfeeding patients
* Patients responding to a contraindication to performing an MRI
* Patient under state medical aid (AME)
* Adult patients protected by law

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2016 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2030-03-15 (Estimated); Study Completion 2030-03-15 (Estimated)

PRIMARY OUTCOMES:
Image quality | 7 years
  The main evaluation criterion will be the choice of the two (or three) evaluators as to the best sequence between the new sequence and the standard sequence.

SECONDARY OUTCOMES:
Acquisition period | 7 years
  Average acquisition time
Apnea | 7 years
  Proportion of patients for whom apnea was requested.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté LEWIN, MD, PHD, Principal Investigator — APHP
Locations (1):
- CHU Paul Brousse, Villejuif, France

IPD SHARING:
Plan to Share IPD: No